CLINICAL TRIAL: NCT04794114
Title: enGIneering For sporT for All
Acronym: GIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 713
Record Dates: First submitted 2021-02-11; First posted 2021-03-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
Keywords: orthosis; hemiplegia
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- orthosis in hemiplegia (Experimental)
  Interventions: Device: experimental ankle foot orthosis; Device: traditional ankle foot orthosis

INTERVENTIONS:
Device: experimental ankle foot orthosis — On the basis of an accurate kinetic and kinematic analysis, a customized orthosis in thermoplastic material with carbon inserts will be created that will make the brace more elastic and facilitate the child's motor activities.
Device: traditional ankle foot orthosis — The normal afos in thermoplastic material, while guaranteeing an ankle joint stability, make the joint more rigid and reduce the elasticity of movement especially during running, jumping and sprinting.

SUMMARY:
hemiplegia is a pathological condition that affects one side of the body which is associated with difficulty in maintaining an upright posture and walking and which is commonly compensated for by using orthoses (AFO). However, the orthoses are inadequate for sports from a design and prescription point of view, which specifies that the goal of the orthosis is to support walking and that any other use compromises its reliability.

The main objective therefore provides for an improvement in the involvement of these children in sports activities (both at school and during leisure time) through the development of new generation orthoses.

DETAILED DESCRIPTION:
The main objective therefore provides for an improvement in the involvement of these children in sports activities (both at school and during leisure time) through the development of new generation orthoses.

Secondary objective: the second objective involves the verification of the orthosis previously designed and built, ie the device must comply with the project specifications and allow the patient to perform sports activities. Correct functioning will be tested by functional evaluation of the model developed through biomechanical analysis of movement performed indoors (in the laboratory) and outdoors.

Notes on the calculation of the sample size: the project foresees the involvement at the moment of 20 children with hemiplegia under treatment at MEDEA to whom an overall improvement of the living conditions is to be guaranteed.

Steps: 1-Technology design - "to play together" 2 - Analysis and identification of the guidelines for the prescription of use; 3 - Evaluation of the motor biomechanical situation of subjects wearing orthoses: indoor and outdoor to evaluate the limits of the orthosis used; 4 - identification of indicators for the evaluation of motor performance; 5 - Identification of the technical specifications (functional and clinical, mechanical, structural, geometric, materials, design) of the new generation orthosis-sensor system.

6- Definition of inclusion criteria, recruitment of 20 subjects starting from Medea and contacts with schools and families to which they belong.

7- Validation- "to verify it really runs" WP5.1 - Functional evaluation of the model developed through biomechanical analysis of movement carried out in the laboratory.

The I.R.C.C.S E. Medea will appropriately select 20 children with hemiplegia and wearers of orthoses.

A biomechanical assessment will be performed through gait analysis to identify the limits of the orthosis used.

8- Two conditions will be evaluated:

* walking tests without orthoses;
* walking tests with orthoses usually used. From the comparative analysis of the collected data, the criticalities of the device will be defined in order to identify the project specifications of the new generation orthosis.

  9-Following the design and construction of the new AFO, a biomechanical evaluation will be performed again by means of gait analysis to validate its correct functioning.

  10- Further validation will be performed using virtual reality environments (GRAIL Gait Real time Analysis Interactive Lab).

After a rehabilitation process, once a certain degree of confidence has been reached in the use of the new orthosis, the device will be tested using outdoor wearable sensors. By doing so, it will be possible to identify indicators for the evaluation of sports performance.

ELIGIBILITY:
Inclusion Criteria:

* Users of Ankle Foot Orthosis (AFO) without any time limit;
* GMFCS 1-2 scale values;
* Ashworth triceps sural values <= 3.

Exclusion Criteria:

* patients using knee and hip orthoses (KAFO, HKAFO);
* patients who need assisted walking (use of crutches, walkers or other);
* uncooperative patients.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
gait analysis with standard ankle foot orthosis | The evaluations are performed before the new ankle foot orthosis is delivered
  kinematic (joint angle during gait cycle) and kinetic evaluation (power generation and absorption and moments) both with standard orthosis
gait analysis with experimental ankle foot orthosis | The evaluations are performed 1 month after the new ankle foot orthosis is delivered
  kinematic (joint angle during gait cycle) and kinetic evaluation (power generation and absorption and moments) both with experimental orthosis

SECONDARY OUTCOMES:
G- sensor with standard ankle foot orthosis | The evaluations are performed before the new ankle foot orthosis is delivered
  accelerometric evaluation during running and sprinting (linar parameters, velocity, step length, cadency) with standard orthosis
G- sensor with experimental ankle foot orthosis | The evaluation is performed 1 month after the new ankle foot orthosis is delivered
  accelerometric evaluation during running and sprinting (linar parameters, velocity, step length, cadency) with experimental orthosis

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No